CLINICAL TRIAL: NCT04606771
Title: A Multi-centre Phase II, Double-Blind, Randomised Study of Savolitinib in Combination With Osimertinib vs Savolitinib in Combination With Placebo in Patients With EGFRm+ and MET Amplified Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Progressed Following Treatment With Osimertinib
Brief Title: A Study Comparing Savolitinib Plus Osimertinib vs Savolitinib Plus Placebo in Patients With EGFRm+ and MET Amplified Advanced NSCLC
Acronym: CoC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5084C00009
Record Dates: First submitted 2020-09-01; First posted 2020-10-28 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally; Advanced; Metastatic; Carcinoma; Non-Small Cell Lung Cancer; Osimertinib; Tagrisso; Savolitinib; MET; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Carcinoma | interventions — osimertinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Intervention Model Description: 1. Patients will take savolitinib 300mg tablets QD within 15 minutes after the start of a meal except for the day on which PK samples are taken. Patients will take osimertinib 80mg tablet once daily with/without food except for the day on which PK samples are taken. On the day when PK samples are taken both savolitinib & osimertinib will be administered after a meal prepared by the clinic
  2. Patients will take savolitinib 300mg tablets QD within 15 minutes after the start of a meal except for the day on which PK samples are taken. Patients will take placebo to osimertinib 80mg tablet once daily with/without food except for the day on which PK samples are taken. On the day when PK samples are taken both savolitinib & placebo to osimertinib will be administered within 15 minutes after a meal prepared by the clinic
  In addition to comparing the ORR between groups, this study will also assess safety and tolerability, DoR, DCR, OS, PFS and other measures of antitumor activity
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Savolitinib 300 mg oral QD
  Osimertinib 80 mg oral QD
  Interventions: Drug: Osimertinib + Savolitinib
- Arm B (Experimental): Savolitinib 300 mg oral QD
  Placebo to Osimertinib 80mg oral QD
  Interventions: Drug: Savolitinib + Placebo

INTERVENTIONS:
Drug: Osimertinib + Savolitinib — Osimertinib 80 mg oral QD
  Savolitinib 300mg oral QD
  Arms: Arm A
Drug: Savolitinib + Placebo — Savolitinib 300mg Oral QD
  Placebo to Osimertinib 80mg oral QD
  Arms: Arm B

SUMMARY:
This study will compare the activity of the combination of savolitinib and osimertinib against the combination of savolitinib with placebo to osimertinib in patients with Epidermal Growth Factor Receptor Mutation Positive and MET amplified, locally advanced or metastatic non-small cell lung cancer who have progressed following treatment with osimertinib.

DETAILED DESCRIPTION:
Resistance to EGFR-TKIs is a clinical problem. One of the mechanisms for resistance to osimertinib is amplification of the MET receptor tyrosine kinase, which activates downstream intracellular signalling independent of EGFR. This study will explore the individual contribution of savolitinib to MET mediated osimertinib resistance, by assessing the response to dual pathway blockade of EGFRm and MET to overcome MET mediated resistance to osimertinib versus inhibition of the MET pathway alone by investigating the efficacy of savolitinib plus osimertinib versus savolitinib plus placebo to osimertinib (hereafter referred to as placebo) in patients with EGFRm+ and MET amplified, locally advanced or metastatic NSCLC who have progressed following treatment with osimertinib. This is a multi centre, Phase II, double blind, randomised study.

Patients will be randomised in a ratio of 1:1 to receive treatment with savolitinib once daily plus osimertinib once daily or savolitinib once daily plus placebo. Randomisation will be stratified according to the number ofprior lines of therapy (ie, osimertinib monotherapy as first line or ≥ second line [which includes patients who received osimertinib monotherapy before or after chemotherapy]). All patients confirmed as eligible will begin treatment on Day 1 with savolitinib plus osimertinib or savolitinib plus placebo. Treatment will continue once daily in 28 day cycles until either objective PD by RECIST 1.1 is assessed, unacceptable toxicity occurs, consent is withdrawn, or another discontinuation criterion is met.

After progression, patients can be unblinded, and patients initially randomised to the savolitinib plus placebo arm may cross-over to open-label savolitinib plus osimertinib following investigator assessed objective PD to ensure that all patients enrolled may have the opportunity to receive the combination of savolitinib plus osimertinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age at the time of signing the informed consent (≥ 20 years of age in Japan). All genders are permitted
* Histologically or cytologically confirmed locally advanced or metastatic EGFRm+ NSCLC harbouring an EGFR mutation known to be associated with EGFR TKI sensitivity and that is permitted in the osimertinib national label (such as exon 19 deletion and/or L858R), which is not amenable to curative therapy.
* Documented radiologic PD following treatment with osimertinib (osimertinib does not need to be the most recent therapy).
* Have MET amplification as determined by central MET FISH testing on tumour specimen collected following progression on prior osimertinib treatment.
* At least measurable target lesion
* Patients must have received at least one but no more than 3 prior lines of therapy (including investigational therapy) in the locally advanced/metastatic setting.
* Adequate haematological, liver and renal function
* Eastern Cooperative Oncology Group/WHO performance status of 0 or 1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* Females of childbearing potential should be willing to use adequate contraceptive measures, should not be breastfeeding, and must have a negative pregnancy test.
* Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 6 months following discontinuation of study intervention. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing study intervention.

Exclusion Criteria:

* Unresolved toxicities from any prior therapy greater than CTCAE Grade 1 at the time of starting study intervention with the exception of alopecia, haemoglobin ≥ 9 g/dL and Grade 2, prior platinum therapy related neuropathy.
* As judged by the investigator, active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy.
* Any of the following cardiac diseases currently or within the last 6 months:

  * Unstable angina pectoris
  * Congestive heart failure (NYHA Grade ≥ 2)
  * Acute myocardial infarction
  * Stroke or transient ischemic attack
  * Uncontrolled hypertension (BP ≥ 150/95 mmHg despite medical therapy).
  * Mean resting corrected QT interval (QTcF) > 470 msec for women and > 450 msec for men at Screening, obtained from 3 ECGs using the screening clinic ECG machine derived QTcF value.
  * Any factors that may increase the risk of QTcF prolongation or risk of arrhythmic events
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECGs.
  * Acute coronary syndrome
* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤ 28 days or limited field radiation for palliation ≤ 7 days prior to starting study intervention or has not recovered from side effects of such therapy.
* Major surgical procedures ≤ 28 days of beginning study intervention or minor surgical procedures ≤ 7 days. No waiting is required following port-a-cath placement.
* As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including renal transplant or active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to enter the study or which would jeopardise compliance with the CSP.
* Active HBV (positive HBsAg result) or HCV. Viral testing is not required for assessment of eligibility for the study.
* Known serious active infection including, but not limited to, tuberculosis, or HIV (positive HIV 1/2 antibodies). Testing is not required for assessment of eligibility for the study.
* Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
* Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 2 weeks prior to start of study intervention.
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis, which required steroid treatment, or any evidence of clinically active ILD.
* Prior or current treatment with a 3rd generation EGFR-TKI other than osimertinib.
* Prior or current treatment with savolitinib or another MET inhibitor (for example, foretinib, crizotinib, cabozantinib, onartuzumab, capmatinib).
* Patients who have received ≥ 4 lines of systemic therapy for NSCLC
* Any cytotoxic chemotherapy, investigational agents or other anti cancer drugs for the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days prior to the first dose of study intervention with the exception of monotherapy osimertinib which may continue uninterrupted during screening.
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study intervention) medications or herbal supplements known to be strong inducers of CYP3A4 or strong inhibitors of CYP1A2, or CYP3A4 substrates which have a narrow therapeutic range within 2 weeks of the first dose of study intervention (3 weeks for St John's Wort) will be excluded. All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4 during the study and for 3 months later the last dose intake.
* Participation in another clinical study with a cytotoxic, investigational product, or other anti cancer drug for the treatment of advanced NSCLC if received study intervention from that study within 14 days of the first dose of study intervention.
* Known hypersensitivity to the active or inactive excipients of osimertinib or savolitinib or drugs with a similar chemical structure or class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2026-03-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (2):
  - Research Site, Duarte, California
  - Research Site, Sacramento, California
- Research Site, Buenos Aires, Argentina
- India (2):
  - Research Site, Delhi
  - Research Site, Mumbai
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
  For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5084C00009&attachmentIdentifier=11272ce8-3fc2-4e0a-8bcf-35ba59653ca5&fileName=Clinical_Study_Report_Synopsis-redacted.pdf&versionIdentifier=
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5084C00009&attachmentIdentifier=b033ae41-e281-4c1a-8461-e3e0412b761d&fileName=Protocol_Redacted.pdf&versionIdentifier=
- See also: SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5084C00009&attachmentIdentifier=3acf2019-583a-426e-b6ba-934b962165cf&fileName=Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Savolitinib Plus Osimertinib: Savolitinib 300 mg oral QD
  Osimertinib 80 mg oral QD
- Savolitinib Plus Placebo: Savolitinib 300 mg oral QD
  Placebo to Osimertinib 80mg oral QD
Period: Overall Study
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Started | 14 | 16
Completed | 0 | 0
Not Completed | 14 | 16
Not completed — Patients ongoing study at data cut-off | 9 | 9
Not completed — Death | 5 | 6
Not completed — Wrong randomisation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (11.42) | 62.5 (10.02) | 59.6 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 12 | 15 | 27
  White | 1 | 0 | 1
  Other | 0 | 1 | 1
  Not reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Percentage of evaluable patients with an Investigator-assessed visit response of complete response (CR) or partial response (PR). CR defined as disappearance of all target and non-target lesions and no new lesions. PR defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesions. Overall Response (OR) = CR + PR.
Time Frame: Tumour assessments every 6 weeks from randomisation up to 24 weeks, then every 8 weeks until objective disease progression (maximum of approximately 25 months)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 14 | 16
Percentage of participants | 57.1 [28.86 to 82.34] | 12.5 [1.55 to 38.35]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomised therapy or receives another anti-cancer therapy prior to progression. Progression (i.e., PD) is defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of ≥5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 14 | 16
Months | 7.36 [5.55 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | 1.64 [1.28 to 4.07]

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date of first documented response until date of documented progression per RECIST 1.1 as assessed by the investigator or death in the absence of disease progression.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 8 | 2
Weeks | 30.57 [18.86 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | NA [12.43 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events

4. Secondary Outcome: Tumour Size Assessment (TSA)
Description: TSA is defined as the percentage change from baseline in TLs at 12 weeks per RECIST 1.1 as assessed by the investigator.
Time Frame: Baseline and 12 weeks.
Population: Patients with either a tumour size recorded at 12 weeks or enough information to impute a value.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 12 | 13
Percentage change | -35.0 (29.62) | 8.5 (38.95)

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomisation until the date of death due to any cause.
Time Frame: From the date of randomisation until death due to any cause, assessed up to the data cut-off date (21 December 2022) (maximum of approximately 25 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 14 | 16
Months | NA [9.56 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events | 13.37 [7.82 to NA] — NA - Not calculated, estimates cannot be calculated due to too few events

6. Secondary Outcome: Total Clearance in EGFR Mutations at 6-weeks After Therapy Initiation (Percentage Change From Baseline in EGFR Mutation Allele Frequencies).
Description: To determine the prevalence of ctDNA clearance after savolitinib plus osimertinib or savolitinib plus placebo treatment in this patient population
Time Frame: 6-weeks after therapy initiation.
Measure: Mean (Standard Deviation); unit: Allele Frequency
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 3 | 8
Allele Frequency | -93.6 (11.03) | -62.7 (48.73)

7. Secondary Outcome: Total Clearance in EGFR Mutations at 6-weeks After Therapy Initiation (Absolute Change From Baseline in EGFR Mutation Allele Frequencies).
Description: as for outcome 6
Time Frame: 6-weeks after therapy initiation.
Measure: Mean (Standard Deviation); unit: Allele Frequency
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 3 | 8
Allele Frequency | -17.4 (17.59) | -2.9 (2.93)

8. Secondary Outcome: PK Concentration Ratios on Multiple Dosing
Description: The time dependency of the PK on multiple dosing is assessed by the ratio of mean concentrations at the timepoints identified in column one. For example, the Geometric mean ratio for "C3h Cycle2 Day 1 / C3h Cycle 1 Day 1" periods is the geometric mean value for C3h Cycle 2 Day 1 (Stage 2) divided by the geometric mean value for C3h Cycle 1 Day 1 (Stage 1). Because the measurement is a ratio of values, no measures of central tendency are appropriate.
Time Frame: C3h Cycle 2 Day 1/C3h Cycle 1 Day 1; Cpre-dose Cycle 3 Day 1/Cpre-dose Cycle 2 Day 1; Cpre-dose Cycle 6 Day 1/Cpre-dose Cycle 2 Day 1; Cpre-dose Cycle 11 Day 1/Cpre-dose Cycle 2 Day 1. (Each Cycle is 28 days)
Population: Geometric mean ratios provided for three different visit combinations
Measure: Number; unit: Geometric mean ratio
Groups:
- Savolitinib: Savolitinib 300 mg oral QD
- Osimertinib: Osimertinib 80mg oral QD
Arm/Group | Savolitinib | Osimertinib
Number analyzed (Participants) | 30 | 14
Geometric mean ratio
  C3h Cycle 2 Day 1 / C3h Cycle 1 Day 1 | 0.8812 | 1.081
  Cpre-dose Cycle 3 Day 1 / Cpre-dose Cycle 2 Day 1 | 0.8650 | 1.032
  Cpre-dose Cycle 6 Day 1 / Cpre-dose Cycle 2 Day 1 | 0.6352 | 1.068

9. Secondary Outcome: AUCss of Savolitinib, Osimertinib and Their Metabolites, (M2 and M3 for Savolitinib; AZ5104 for Osimertinib)
Description: Area under the plasma concentration-time curve at steady state
Time Frame: Cycle 3, Day 1: Pre-dose and 1, 3, 4, and 6 hours post-dose
Population: All patients with PK data are analysed for savolitinib, osimertinib and their metabolites
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 13 | 5
h*ng/mL
  Savolitinib | 7875 (37.54) | 11890 (37.56)
  M2 | 2630 (48.80) | 3516 (44.43)
  M3: number analyzed (Participants) | 12 | 5
  M3 | 966.7 (49.07) | 1348 (42.37)
  Osimertinib: number analyzed (Participants) | 13 | 0
  Osimertinib | 12910 (50.80) |
  AZ5104: number analyzed (Participants) | 13 | 0
  AZ5104 | 1086 (70.80) |

10. Secondary Outcome: Cssmax of Savolitinib, Osimertinib and Their Metabolites, (M2 and M3 for Savolitinib; AZ5104 for Osimertinib)
Description: Maximum steady state plasma concentration
Time Frame: Cycle 3, Day 1: Pre-dose and 1, 3, 4, and 6 hours post-dose
Population: All patients with PK data are analysed for savolitinib, osimertinib and their metabolites
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 13 | 7
ng/mL
  Savolitinib | 1282 (35.65) | 2058 (32.00)
  M2 | 351.0 (39.91) | 581.5 (21.19)
  M3 | 129.0 (34.90) | 213.9 (36.08)
  Osimertinib: number analyzed (Participants) | 13 | 0
  Osimertinib | 678.3 (50.80) |
  AZ5104: number analyzed (Participants) | 13 | 0
  AZ5104 | 51.23 (70.14) |

11. Secondary Outcome: Tssmax of Savolitinib, Osimertinib and Their Metabolites, (M2 and M3 for Savolitinib; AZ5104 for Osimertinib)
Description: Time to maximum plasma concentration at steady state
Time Frame: Cycle 3, Day 1: Pre-dose and 1, 3, 4, and 6 hours post-dose
Population: All patients with PK data are analysed for savolitinib, osimertinib and their metabolites
Measure: Median (Full Range); unit: h
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 13 | 7
h
  Savolitinib | 3.00 [1.00 to 5.62] | 3.00 [0.95 to 6.00]
  M2 | 3.00 [1.00 to 5.62] | 1.05 [0.95 to 6.00]
  M3 | 3.00 [0.92 to 5.78] | 1.05 [0.95 to 6.00]
  Osimertinib: number analyzed (Participants) | 13 | 0
  Osimertinib | 4.00 [3.00 to 6.00] |
  AZ5104: number analyzed (Participants) | 13 | 0
  AZ5104 | 4.00 [0.00 to 6.00] |

12. Secondary Outcome: CLss/F of Savolitinib, Osimertinib and Their Metabolites, (M2 and M3 for Savolitinib; AZ5104 for Osimertinib)
Description: To evaluate the PK of savolitinib and osimertinib.
Time Frame: Cycle 3, Day 1 (Each Cycle is 28 days)
Population: All patients with PK data are analysed for savolitinib, osimertinib and their metabolites
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
Number analyzed (Participants) | 13 | 5
L/h
  Savolitinib | 38.10 (37.54) | 25.23 (37.56)
  M2 | 114.1 (48.80) | 85.32 (44.43)
  M3: number analyzed (Participants) | 12 | 5
  M3 | 310.3 (49.07) | 222.5 (42.37)
  Osimertinib: number analyzed (Participants) | 13 | 0
  Osimertinib | 0.01241 (50.80) |
  AZ5104: number analyzed (Participants) | 13 | 0
  AZ5104 | 0.1475 (70.80) |

ADVERSE EVENTS:
Time Frame: Collected throughout the study, from date of informed consent until 28 days after the last dose of study treatment (or end of follow up period). All-cause mortality (death due to any cause): from randomisation up to data cut-off date (21 Dec 2022). Maximum timeframe of approximately 24.4 months.
Arm/Group | Savolitinib Plus Osimertinib | Savolitinib Plus Placebo
All-Cause Mortality (participants affected / at risk) | 5/14 | 7/16
Serious Adverse Events (participants affected / at risk) | 4/14 | 3/16
Other Adverse Events (participants affected / at risk) | 13/14 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Savolitinib Plus Osimertinib (N=14) | Savolitinib Plus Placebo (N=16)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Savolitinib Plus Osimertinib (N=14) | Savolitinib Plus Placebo (N=16)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 5 (6) | 4 (4)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 2 (2) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 2 (3) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT04606771/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT04606771/SAP_001.pdf